CLINICAL TRIAL: NCT05975359
Title: A Pilot Study of the Interi Manifold With Traditional Surgical Drains in Implant-Based Breast Reconstruction
Brief Title: Assessment of the Interi Manifold in Implant-Based Breast Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: IC Surgical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-69609; NCI-2024-02053 (Registry Identifier: National Cancer Institute Clinical Trials Reporting Program)
Record Dates: First submitted 2023-07-27; First posted 2023-08-03 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Mastectomy; Implant Based Breast Reconstruction

STUDY DESIGN:
Intervention Model Description: Patients undergoing bilateral mastectomy will be eligible for this study. Each patient will receive both the Interi manifold (intervention arm) and the JP drain (comparison arm) placed in different breasts. Drain placement will be simultaneous. The laterality of different drain systems (intervention and comparison study arms) will be randomly assigned for each patient.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Interi Manifold Drain System (Experimental): Following bilateral mastectomy, stage 1 surgery for immediate implant-based breast reconstruction will be performed in each patient breast. The breast randomized to treatment with the Interi manifold (intervention arm) will have the Interi manifold placed alongside the tissue expander intra-operatively. Surgical reconstruction, closure, and post-operative management will proceed as standard. Postoperative follow-up will occur within 1 week of surgery. Weekly follow-ups with documentation of clinical data throughout recovery will also take place until removal of the Interi drain system, which typically occurs 1-3 weeks after surgery. Criteria for drain removal is defined as 2 consecutive days with drain output below 30 mL. While drains are in place, patients will be required to monitor drain output and keep a daily drain log.
  Interventions: Device: Interi Manifold Drain System
- Jackson Pratt Drain System (Active Comparator): Following bilateral mastectomy, stage 1 surgery for immediate implant-based breast reconstruction will be performed in each patient breast. The breast randomized to treatment with the Jackson Pratt drain (active comparator arm) will have the Jackson Pratt drain placed alongside the tissue expander intra-operatively. Surgical reconstruction, closure, and post-operative management will proceed as standard. Postoperative follow-up will occur within 1 week of surgery. Weekly follow-ups with documentation of clinical data throughout recovery will also take place until removal of the Jackson Pratt drain system, which typically occurs 1-3 weeks after surgery. Criteria for drain removal is defined as 2 consecutive days with drain output below 30 mL. While drains are in place, patients will be required to monitor drain output and keep a daily drain log.
  Interventions: Device: Jackson Pratt Drain System

INTERVENTIONS:
Device: Interi Manifold Drain System — The Interi manifold surgical drain system will be placed in the breast pocket during stage 1 immediate implant based breast reconstruction. Output of the interi drain will be monitored daily and the Interi drain will remain in the surgical site until criteria for drain removal are met. Removal of the Interi drain will be performed in clinic by surgical staff.
  Other Names: Interi manifold; Interi drain; Interi surgical drain
  Arms: Interi Manifold Drain System
Device: Jackson Pratt Drain System — The Jackson Pratt surgical drain system will be placed in the breast pocket during stage 1 immediate implant based breast reconstruction. Output of the Jackson Pratt drain will be monitored daily and the drain will remain in the surgical site until criteria for drain removal are met. Removal of the Jackson Pratt drain will be performed in clinic by surgical staff.
  Other Names: JP drain; JP surgical drain
  Arms: Jackson Pratt Drain System

SUMMARY:
Patients with breast cancer that elect to undergo implant-based breast reconstruction (IBBR) often require the placement of a surgical drain. Surgical drains are used to manage dead space and prevent seroma formation or accumulation of fluid within the surgical field postoperatively. The most frequently used drain is a Jackson-Pratt (JP) drain, which is limited by poor surgical site coverage and low capacity, leading to inconsistent suction and prolonged time that a drain is left in place. The Interi Drain system is a novel, multi-branched manifold with a proprietary suction system that provides consistent suction and addresses many of the shortcoming of JP drains. The purpose of this study is to compare the Interi system to standard JP drains across outcomes including number of surgical drain sites, complication rates, time to drain removal, time to initiate tissue expansion, total fluid volume drained, and patient satisfaction.

DETAILED DESCRIPTION:
Patients seeking a mastectomy with immediate tissue expander/implant-based breast reconstruction will be considered. Potential participants will be screened for inclusion and exclusion criteria and informed of the study protocols, risk, and potential benefits.

Consenting patients who meet eligibility criteria will undergo bilateral mastectomy and immediate, implant-based breast reconstruction using a tissue expander. On the day of surgery, patient breasts will be randomized into the Interi cohort or the JP cohort, such that in each patient one breast receives the Interi drain and the other receives JP drains. Randomization will be stratified by the laterality of the primary tumor. The respective drains will be placed intraoperatively.

Postoperative care will proceed as standard. Postoperative follow-up will occur within 1 week of surgery. Weekly follow-ups with documentation of clinical data throughout recovery will also take place until removal of the drain systems, which typically occurs 1-3 weeks after surgery. While drains are in place, patients will be required to monitor drain output and keep a daily drain log. Thereafter, follow-ups will be scheduled as needed (monthly) according to the usual clinical practice of implant-based breast reconstruction. This will include routine tissue expansion in preparation for the second stage expander to definitive implant exchange.

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer diagnosis (any form) or Genetic mutation with presence of breast mass.
2. Indication for bilateral mastectomy
3. Plan for immediate, implant-based pre-pectoral breast reconstruction using an acellular dermal matrix
4. Age 18 - 65
5. Female Sex
6. Ability to understand and the willingness to personally sign the written IRB-approved informed consent document (English language).

Exclusion Criteria:

1. Have a prior history of radiation to the breast or planned radiotherapy to the breast within the first year post-operatively.
2. Are enrolled in another study that requires the concomitant use of any investigational product during the study period that the Principal Investigator believes will interfere with study endpoints.
3. Have received oncologic chemotherapy within the past 21 days or planned within the time fame of the study intervention. Have received antiplatelet therapy (other than aspirin) and/ or other anticoagulation therapy in the past 60 days.
4. Are a smoker or use illicit drugs.
5. Any prior allergic reaction to Teflon.
6. Are pregnant or nursing.
7. Are undergoing a delayed reconstruction following mastectomy.
8. HIV infection, active UTI infection, or other active infection.
9. Those requiring more than one Manifold for fluid removal per breast will be excluded.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Device safety | Complications will be recorded until stage 2 surgery (replacement of tissue expanders with permanent implants), which typically occurs after 6 months.
  Incidence of adverse events or complications (e.g. seroma, hematoma, infection, dehiscence, etc.) will be recorded for both drain systems.
Time to drain removal | Drain removal typically occurs between 1-3 weeks post-op.
  The number of days between placement of each drain system (stage 1 surgery) and removal of the drain (defined as 2 consecutive days with drain output below 30 mL).

SECONDARY OUTCOMES:
Number of drain sites | This will be recorded by the surgeon immediately after completion of the stage 1 operation.
  The number of drain sites (holes exiting the surgical site) in each breast.
Total fluid drained | Drain removal typically occurs between 1-3 weeks post-op.
  The amount of fluid (mL) collected by each surgical drain from the operative breast for the duration of drain placement will be recorded for both drain systems.
Time to initiate tissue expansion | Tissue expansion typically begins 3-6 weeks after stage 1 surgery.
  The amount of time in days after tissue expander placement (same operative time point as drain placement) for a patient to begin tissue expansion (when determined clinically appropriate by the attending physician).
Patient satisfaction (BreastQ) | Administration of BreastQ will occur at specific post-operative time points (e.g. 1 week, 3 weeks, 6 months, and 1 year).
  Both quality of life and patient satisfaction will be assessed by validated patient survey (BreastQ). Each breast will be assessed independently by the patient to determine if the type of drain has affected the patient's perception of their recovery.
Patient satisfaction (study-specific survey) | Administration of the study specific survey will occur at specific post-operative time points (e.g. 1 week, 2 weeks, and at drain removal).
  Patient satisfaction with each drain system and ease of use will be assessed using a study-specific survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Hospital and Clinics, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No